CLINICAL TRIAL: NCT07297173
Title: Phase 1 Study of Chemotherapy Combining With HLA-mismatched G-CSF Mobilized Peripheral Blood Mononuclear Cell Infusion as a Bridge to Allogeneic Hematopoietic Stem Cell Transplantation for Relapsed and Refractory Leukemia
Brief Title: Phase 1 Study of Chemotherapy Plus HLA-mismatched GPBMC Infusion Bridging to Allo-HSCT for R/R Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allo-GPBMC to Allo-HSCT
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Relapsed Leukemia; Refractory Leukemia
Keywords: HLA-mismatched GPBMC; allo-HSCT; relapsed leukemia; refractory leukemia
MeSH Terms: conditions — Leukemia | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): This cohort includes patients with relapsed and refractory leukemia. Patients firstly receive chemotherapy per center standard, followed by HLA-mismatched GPBMC infusion. Secondly, patients receive HLA-matched sibling/haploidentical/unrelated HSCT.
  Interventions: Procedure: Chemotherapy; Biological: HLA-mismatched GPBMC infusion; Procedure: Allogeneic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Chemotherapy — Available chemotherapy regimens include but not limited to FLAG (fludarabine, cytarabine, G-CSF), DAV (daunorubicin, cytarabine, venetoclax), IAV (idarubicin, cytarabine, venetoclax), VDCP (vincristine, daunorubicin, cyclophosphamide, prednisone), hyper-CVAD A (cyclophosphamide, vincristine, doxorubicin, dexamethasone), FC (fludarabine and cyclophosphamide), et al.
Biological: HLA-mismatched GPBMC infusion — HLA-mismatched GPBMCs are infused following chemotherapy.
Procedure: Allogeneic Stem Cell Transplantation — Patients receive conditioning including but not limited to fludarabine, cyclophosphamide, antithymocyte globulin (ATG), and total body irradiation (TBI). HLA-matched sibling/haploidentical/unrelated GPBMCs are infused at day 0. Post-transplant cyclophosphamide, tacrolimus/cyclosporin, and mycophenolate mofetil are administered as graft-versus-host disease prophylaxis.

SUMMARY:
This is a Phase 1 clinical study designed to evaluate the safety, tolerability, and preliminary efficacy of chemotherapy combining with HLA-mismatched G-CSF mobilized peripheral blood mononuclear cell (GPBMC) infusion as a bridging therapy to allogeneic hematopoietic stem cell transplantation (allo-HSCT) in patients with relapsed and refractory (R/R) leukemia.

DETAILED DESCRIPTION:
Eligible patients will firstly receive chemotherapy combining with infusion of HLA-mismatched GPBMCs with the aim to reduce leukemia burden. Secondly, they will receive allo-HSCT per protocol. GPBMCs used in the first-step infusion will be derived from a sibling or unrelated donor, and GPBMCs used in the allo-HSCT procedure will be derived from an alternative donor, or the same donor (haploidentical/matched sibling/HLA 9-10 loci matched unrelated) as in the first step. The primary endpoint is the incidence of treatment-related adverse events (AEs) within 100 days post allo-HSCT, including graft-versus-host disease (GVHD), infection, organ dysfunction, and hematological toxicity. Secondary endpoints include overall survival (OS) at 1 and 2 years, progression-free survival (PFS), and graft-versus-host disease-free, relapse-free survival (GRFS).

ELIGIBILITY:
Inclusion Criteria:

* Age >=15 years, male or female, non-limited by race or ethnicity.
* Confirmed diagnosis of R/R leukemia and risk stratification according to the World Health Organization (WHO) 5th edition classification, based on histopathology and cytogenetics.
* Adequate hepatic function including alanine transaminase (ALT) and aspartate aminotransferase (AST )<= 3 × upper limit of normal(ULN), and total bilirubin <= 1.5 × ULN.
* Adequate renal function including serum creatinine <= 2 × ULN or CrCl>= 40mL/min.
* LVEF measured by echocardiogram is within the normal range (LVEF > 50%).
* The subject must have one HLA mismatched donor who is >= 18 years old to provide GPBMCs for the first-step infusion. If this donor is not qualified as an allo-HSCT donor, the subject must also have another donor who is >= 18 years old and qualified as allo-HSCT donor (i.e., matched sibling, 9-10/10 loci matched unrelated, or haploidentical). In addition, the donor voluntarily donates hematopoietic stem cells and signs the consent form. Each subject (or his/her legal representatives) must sign the Informed Consent Form (ICF), indicating that he/she understands the purpose and procedures of research, and is willing to participate in research.
* Donor inclusion criteria: The donor meets the institution's criteria for related peripheral blood hematopoietic stem cell donors. The donor must be able to tolerate the cell separation and collection process, and sign the Informed Consent Form.

Exclusion Criteria:

* Uncontrolled infection or hemorrhage.
* Cardiovascular disease with clinical significance, such as uncontrolled or highly symptomatic cardiac arrhythmias, congestive heart failure, or myocardial infarction within 6 months prior to screening, or New York Heart Association (NYHA) function class 3 (moderate) or class 4 (severe) heart disease.
* Uncontrolled autoimmune disease or requiring immunosuppression treatment.
* History of severe blood infusion reaction.
* Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception.
* Psychiatric disorder or cognitive impairment that in the researcher's judgment would make the subject not likely to adhere to the protocol requirements.
* Major surgery within 4 weeks prior to enrollment.
* Life-threatening illness other than leukemia or uncontrolled intercurrent illness.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Graft-Versus-Host Disease (GVHD) | Measured up to 2 years after the last participant is enrolled
  Including acute GVHD (aGVHD) and chronic GVHD (cGVHD), assessed per international universal criteria (e.g., Glucksberg classification).
Infections | Measured up to 2 years after the last participant is enrolled
  Covering bacterial, viral, fungal infections (e.g., pneumonia, sepsis, cytomegalovirus infection), confirmed based on clinical symptoms, laboratory tests, and etiological evidence.
Hematological Toxicity | Measured up to 2 years after the last participant is enrolled
  Including neutropenia, thrombocytopenia, anemia, etc., graded according to the Common Terminology Criteria for Adverse Events (CTCAE) standards.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Measured up to 4 years after the last participant is enrolled
  Time from the completion of allo-HSCT to disease progression, relapse, or death from any cause.
Graft-Versus-Host Disease-Free, Relapse-Free Survival (GRFS) | Measured up to 4 years after the last participant is enrolled
  Time from the completion of allo-HSCT to the first occurrence of any of the following events: grade 3-4 acute GVHD, chronic GVHD requiring systemic treatment, disease relapse, or death.
Overall Survival (OS) | Measured up to 4 years after the last participant is enrolled
  Time from the completion of allo-HSCT to death from any cause.
Treatment-Related Mortality (TRM) | Measured up to 2 years after the last participant is enrolled
  TRM is defined as the death related to treatment instead of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Cai, MD, Principal Investigator — Department of Hematology, the Fifth Medical Center of Chinese PLA General Hospital
Locations (1):
- Department of Hematology, the Fifth Medical Center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided